CLINICAL TRIAL: NCT05451615
Title: Clinical Efficacy and Safety of Real-world Patients With Refractory Rheumatoid Arthritis (D2TRA) Receiving Abatacept in Combination With a Janus Kinase (JAK) Inhibitor
Brief Title: Efficacy and Safety of Abatacept Combined With JAK Inhibitor for Refractory Rheumatoid Arthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zhenhua Ying, Director, Zhejiang Provincial People's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2022018
Record Dates: First submitted 2022-06-17; First posted 2022-07-11 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Abatacept; Treatment Compliance; Rheumatoid Arthritis
MeSH Terms: conditions — Patient Compliance; Arthritis, Rheumatoid | interventions — Janus Kinase Inhibitors; Abatacept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abatacept (Experimental): D2T RA patients receive Abatacept
  Interventions: Drug: Abatacept
- JAK inhibitor (Experimental): D2T RA patients receive JAKi
  Interventions: Drug: Janus Kinase Inhibitor; Drug: Abatacept

INTERVENTIONS:
Drug: Janus Kinase Inhibitor — One group of D2TRA subjects receive Janus Kinase Inhibitors combine Abatacept treatment, another group of D2TRA subjects receive Abatacept treatment only.
  Arms: JAK inhibitor
Drug: Abatacept — One group of D2TRA subjects receive Janus Kinase Inhibitors combine Abatacept treatment, another group of D2TRA subjects receive Abatacept treatment only.

SUMMARY:
The aim of this study is to observe the clinical efficacy and safety of abatacept combined with JAK inhibitor in the treatment of D2TRA patients

ELIGIBILITY:
Inclusion Criteria:

1. Meet the above diagnostic criteria for refractory rheumatoid arthritis
2. The traditional disease-improving rheumatic drug treatment is ineffective, and the use of two or more biological/targeted disease-improving anti-rheumatic drugs is ineffective, and abatacept combined with a JAK inhibitor is required treated patients

Exclusion Criteria:

1. Patients with tumors, hematological diseases, and other autoimmune diseases
2. Those who have a history of allergies to the drugs selected in this study
3. Those who cannot adhere to abatacept combined with JAK inhibitor therapy, or who have serious adverse reactions and did not complete the observation period prescribed by the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Abatacept Combined With JAK Inhibitor for Refractory Rheumatoid Arthritis | maximum 1 years
  The disease activity score of 28 joints with erythrocyte sedimentation rate (DAS28-ESR ≤ 2.6, remission; 2.6 < DAS28-ESR ≤ 3.2, mild activity; 3.2 < DAS28-ESR ≤ 5.1, moderate activity, and DAS28-ESR > 5.1, severe activity)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse EventsArthritis | maximum 1 years
  Liver and kidney function

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Iglesias M, Khalifian S, Oh BC, Zhang Y, Miller D, Beck S, Brandacher G, Raimondi G. A short course of tofacitinib sustains the immunoregulatory effect of CTLA4-Ig in the presence of inflammatory cytokines and promotes long-term survival of murine cardiac allografts. Am J Transplant. 2021 Aug;21(8):2675-2687. doi: 10.1111/ajt.16456. Epub 2021 Feb 18. PMID 33331121

DOCUMENTS (2):
  • Study Protocol (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT05451615/Prot_000.pdf
  • Informed Consent Form (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT05451615/ICF_001.pdf